CLINICAL TRIAL: NCT04772989
Title: A Phase 1/1b Study to Evaluate the Safety and Tolerability of AB308 in Combination With AB122 in Participants With Advanced Malignancies
Brief Title: A Study to Evaluate AB308 in Combination With AB122 in Participants With Advanced Malignancies
Acronym: ARC-12
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Arcus Biosciences, Inc. (Industry)
Collaborators: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: ARC-12; 2021-005589-16 (EudraCT Number); 2024-511116-25-00 (EU CTIS Number)
Record Dates: First submitted 2021-02-22; First posted 2021-02-26 (Actual); Last update posted 2025-08-28 (Actual); Status verified 2024-09

CONDITIONS: Advanced Solid Tumor; Non Small Cell Lung Cancer (NSCLC); Melanoma; Cervical Cancer; Multiple Myeloma; Lymphoma, Non-Hodgkin; Diffuse Large B Cell Lymphoma (DLBCL); Gastric Cancer; Gastroesophageal Junction Adenocarcinoma; Esophageal Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Melanoma; Uterine Cervical Neoplasms; Multiple Myeloma; Lymphoma, Non-Hodgkin; Lymphoma, Large B-Cell, Diffuse; Stomach Neoplasms; Esophageal Neoplasms | interventions — zimberelimab

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (8):
- Dose Escalation Q3W Cohorts (Experimental): Escalating doses of AB308 in combination with zimberelimab (360 mg) will be given every 3 weeks in participants with advanced malignancies.
  Interventions: Drug: AB308; Drug: Zimberelimab
- Dose Escalation Q4W Cohorts (Experimental): Escalating doses of AB308 in combination with zimberelimab (480 mg) will be given every 4 weeks in participants with advanced malignancies.
  Interventions: Drug: AB308; Drug: Zimberelimab
- Dose Escalation Q6W Cohort (Experimental): Selected dose of AB308 in combination with zimberelimab will be given every 6 weeks in participants with advanced malignancies.
  Interventions: Drug: AB308; Drug: Zimberelimab
- Dose Expansion Cohort 1 (Experimental): AB308 will be given in combination with zimberelimab at 360 mg or 480 mg Q3W or Q4W, respectively, in participants with in participants with locally advanced or metastatic NSCLC.
  Interventions: Drug: AB308; Drug: Zimberelimab
- Dose Expansion Cohort 2 (Experimental): AB308 will be given in combination with zimberelimab at 360 mg or 480 mg Q3W or Q4W, respectively, in participants with melanoma.
  Interventions: Drug: AB308; Drug: Zimberelimab
- Dose Expansion Cohort 3 (Experimental): AB308 will be given in combination with zimberelimab at 360 mg or 480 mg Q3W or Q4W, respectively, in participants with metastatic gastric, or gastroesophageal junction, or esophageal cancer.
  Interventions: Drug: AB308; Drug: Zimberelimab
- Dose Expansion Cohort 4 (Experimental): AB308 will be given in combination with zimberelimab at 360 mg or 480 mg Q3W or Q4W, respectively, in participants with cervical cancer.
  Interventions: Drug: AB308; Drug: Zimberelimab
- Dose Expansion Cohort 5 (Experimental): AB308 will be given in combination with zimberelimab at 360 mg or 480 mg Q3W or Q4W, respectively, in participants with hematological malignancies.
  Interventions: Drug: AB308; Drug: Zimberelimab

INTERVENTIONS:
Drug: AB308 — Administered intravenously (IV) as specified in the treatment arm
Drug: Zimberelimab — Administered IV as specified in the treatment arm
  Other Names: AB122

SUMMARY:
This is a Phase 1/1b, multicenter, open-label, dose-escalation, and dose-expansion study to evaluate the safety, tolerability, pharmacokinetic (PK), pharmacodynamic (PD), and clinical activity of AB308 in combination with zimberelimab (AB122) in participants with advanced malignancies.

ELIGIBILITY:
Inclusion Criteria:

* Capable of giving signed informed consent, which includes compliance with the requirements and restrictions listed in the informed consent form (ICF) and in this protocol.
* Male or female participants ≥ 18 years of age (or age ≥ regionally approved age of consent for participation in investigational clinical studies) at the time of signing the informed consent.
* Contraceptive use by men and women should be consistent with local regulations regarding the methods of contraception for those participating in clinical studies.
* Eastern Cooperative Oncology Group (ECOG) performance status score of 0 or 1
* Adequate organ and marrow function

Exclusion Criteria:

* History of trauma or major surgery within 28 days prior to the first dose of study treatment.
* Prior treatment with an anti-TIGIT antibody.
* Any active or prior autoimmune disease that required treatment within 3 years of the first dose of study treatment.
* Prior chemotherapy, targeted small-molecule therapy, immunotherapy, or biologic agents, or use of other investigational drugs within 28 days before first dose of study treatment.
* Discontinued prior immunotherapy for immune related adverse events with a high severity.

NOTE: Other protocol defined Inclusion/Exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 94 (Actual)
Dates: Start 2021-03-19 (Actual); Primary Completion 2025-08-25 (Actual); Study Completion 2025-08-25 (Actual)

PRIMARY OUTCOMES:
Percentage of participants with Adverse Events | From first study treatment administration until up to 90 days after the last dose (Approximately 1 year)
Percentage of participants who experience a Dose Limiting Toxicity | From first study treatment administration through Day 21 (Q3W arm) or Day 28 (Q4W arm) or Day 42 (Q6W arm)

SECONDARY OUTCOMES:
Serum concentration of AB308 | Recorded at baseline (day 1 of cycle 1), during each of the first 5 cycles (each cycle is 21 days or 28 days or 42 days) and up to the first 16 cycles of treatment (up to 22 months), and 30 and 90 days post last dose (up to approximately 25 months)
Serum concentration of zimberelimab | Recorded at baseline (day 1 of cycle 1), during each of the first 5 cycles (each cycle is 21 days or 28 days or 42 days) and up to the first 16 cycles of treatment (up to 22 months), and 30 and 90 days post last dose (up to approximately 25 months)
Percentage of participants with anti-drug antibodies to AB308 | Recorded at baseline (day 1 of cycle 1), during each of the first 5 cycles (each cycle is 21 days or 28 days or 42 days) and up to the first 16 cycles of treatment (up to 22 months), and 30 and 90 days post last dose (up to approximately 25 months)
Percentage of participants with anti-drug antibodies to zimberelimab | Recorded at baseline (day 1 of cycle 1), during each of the first 5 cycles (each cycle is 21 days or 28 days or 42 days) and up to the first 16 cycles of treatment (up to 22 months), and 30 and 90 days post last dose (up to approximately 25 months)
Percentage of participants with Objective Response | From study enrollment until participant discontinuation, first occurrence of progressive disease, or death from any cause, whichever occurs first (up to approximately 3-5 years)
Duration of Response | From the date of first occurrence of a documented objective response to first documentation of disease progression or death from any cause, whichever occurs first (up to approximately 3-5 years)
Percentage of Participants with Disease Control (complete response, partial response, or stable disease) for >6 months | From study enrollment until disease progression or loss of clinical benefit (up to approximately 3-5 years)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Arcus Biosciences
Locations (22):
- United States (15):
  - UCLA Department of Medicine - Hematology/Oncology, Los Angeles, California
  - Mayo Clinic Jacksonville - PPDS, Jacksonville, Florida
  - Goshen Health System, Goshen, Indiana
  - Holden Comprehensive Cancer Center, Iowa City, Iowa
  - Norton Cancer Insititute-Downtown, Louisville, Kentucky
  - Mayo Clinic Rochester, Rochester, Minnesota
  - Columbia University Medical Center, New York, New York
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - University of Oklahoma Peggy and Charles Stephenson Cancer Center, Oklahoma City, Oklahoma
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - Tennessee Onocology - Nashville, Nashville, Tennessee
  - START South Texas Accelerated Research Therapeutics, San Antonio, Texas
  - START South Texas Accelerated Research Therapeutics - Mountain Region, West Valley City, Utah
  - Virginia Cancer Specialists, Fairfax, Virginia
  - University of Wisconsin - Madison, Madison, Wisconsin
- Poland (2):
  - Specjalistyczna Praktyka Lekarska Slawomir Mandziuk, Lubin
  - Med-Polonia Sp. z o.o., Poznan
- Spain (5):
  - Hospital Universitario Vall d'Hebron, Barcelona
  - Clínica Universidad de Navarra - Madrid, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
  - START MADRID Hospital Unviersitario Fundacion Jimenez Diaz, Madrid
  - Clínica Universidad de Navarra, Pamplona

IPD SHARING:
Plan to Share IPD: Yes
Arcus will provide access to individual de-identified participant data and related study documents (e.g., protocol, Statistical Analysis Plan [SAP], Clinical Study Report [CSR]) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions.
  For more information, please visit our website.
Supporting Information: Study Protocol, SAP, CSR
URL: https://trials.arcusbio.com/our-transparency-policy

REFERENCES:
- See also: ARC-12 - Public website — https://trials.arcusbio.com/study/?id=ARC-12